CLINICAL TRIAL: NCT00568659
Title: The Specific Lung Elastance in ALI/ARDS Patients in Supine and Prone Position
Brief Title: The Specific Lung Elastance in Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS) Patients in Supine and Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Gas exchange; Respiratory mechanics; Ventilator Induced Lung Injury
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: specific elastance

INTERVENTIONS:
Procedure: specific elastance — The investigators study the specific lung elastance in ALI/ARDS patients in supine and prone position.

SUMMARY:
The investigators aim is to study the specific lung elastance in ALI/ARDS patients during invasive mechanical ventilation, in supine and prone position.

DETAILED DESCRIPTION:
In sedated and paralyzed ALI/ARDS patients, we study and compare the specific lung elastance in supine and prone position during invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* ALI/ARDS patients during invasive mechanical ventilation

Exclusion Criteria:

* Haemodynamic failure, pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2010-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Specific elastance | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy